CLINICAL TRIAL: NCT01338792
Title: A Phase II Trial of Oxaliplatin and Pemetrexed in Hormone Refractory Prostate Cancer
Brief Title: Oxaliplatin and Pemetrexed Disodium in Treating Patients With Refractory Hormone-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4P-05-7; NCI-2011-00500 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-04-15; First posted 2011-04-20 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-02

CONDITIONS: Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Oxaliplatin; Pemetrexed; Reverse Transcriptase Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy and enzyme inhibitor) (Experimental): Patients receive oxaliplatin IV over 2 hours and pemetrexed disodium IV on day 1. Courses repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: oxaliplatin; Drug: pemetrexed disodium; Other: questionnaire administration; Other: laboratory biomarker analysis; Genetic: reverse transcriptase-polymerase chain reaction; Genetic: polymorphism analysis

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: pemetrexed disodium — Given IV
  Other Names: ALIMTA; LY231514; MTA
Other: questionnaire administration — Ancillary studies
Other: laboratory biomarker analysis — Correlative studies
Genetic: reverse transcriptase-polymerase chain reaction — Correlative studies
  Other Names: RT-PCR
Genetic: polymorphism analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving oxaliplatin and pemetrexed disodium together works in treating patients with refractory hormone-resistant prostate cancer. Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving oxaliplatin together with pemetrexed disodium may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the response rate by Response Evaluation Criteria In Solid Tumors (RECIST) criteria, prostate-specific antigen (PSA) response by the PSA Working Group criteria, and overall clinical benefit defined by summation of RECIST complete responses (CR) plus RECIST partial responses (PR) plus PSA PRs. SECONDARY OBJECTIVES: I. To determine time to progression in patients with hormone-refractory prostate cancer (HRPC) receiving oxaliplatin and pemetrexed. II. To describe the safety profile of this treatment. III. Pain response will be evaluated in an exploratory manner. IV. Undertake a pilot analysis of excision repair cross-complementing 1 (ERCC1) expression levels and polymorphisms, looking at their ability to predict response to platinum therapy. OUTLINE: Patients receive oxaliplatin intravenously (IV) over 2 hours and pemetrexed disodium IV on day 1. Courses repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer
* Measurable disease on computed tomography (CT) or evaluable disease on bone scan with an elevated PSA
* For patients who did not initially present with metastatic disease, definitive treatment with either radical prostatectomy or external beam radiation is permitted
* Documented progression on (a) two prior hormone treatments AND (b) one or two chemotherapy regimens
* Documented progression on two prior hormone therapies is defined as orchiectomy followed by anti-adrenal medication upon progression OR gonadotropin-releasing hormone (GnRH) analog +/- androgen receptor blocker with addition or subtraction upon progression; castrate level of testosterone must be documented at study entry
* Documented progression on taxane-based chemotherapy; in addition, patients may have failed a second prior chemotherapy regimen
* Palliative radiation therapy for metastatic disease is allowed only if less than 25% of total body bone marrow was irradiated; 28 days must have elapsed since completion of radiation therapy (RT) with bone marrow recovery; soft tissue disease irradiated in the prior 2 months may not be designated as measurable disease
* ECOG performance score of 0-2
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelet count >= 100,000/uL
* Creatinine clearance >= 45 mL/min
* Serum total bilirubin =<1.5 mg/dL
* Alkaline phosphatase =< 3x the upper limit of normal (ULN) for the reference lab (=< 5x the ULN for patients with known hepatic metastases) and no upper limit for patients with known bone metastases
* Serum glutamic oxaloacetic transaminase (SGOT)/serum glutamic pyruvic transaminase (SGPT) =< 3x the ULN for the reference lab (=< 5x the ULN for patients with known hepatic metastases)
* Patients must be recovered from both acute and late effects of any prior surgery, radiotherapy or other antineoplastic therapy
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial
* Men of childbearing potential must consent to use barrier contraception while on treatment and for 90 days thereafter
* Patients with pleural or peritoneal effusions are eligible
* Willingness and ability to take vitamin supplementation and steroid premedication as specified in protocol
* Patients with superficial bladder cancer or skin cancer who have second malignancy within 5 years which was removed with curative intent

Exclusion Criteria:

* Active infection or with a fever >= 38.5 degrees Celsius (C) within 3 days of the first scheduled protocol treatment
* Patients with brain metastases
* Prior malignancy within the past 5 years, except for curatively treated basal cell or squamous cell carcinoma of the skin or superficial bladder cancer
* Known hypersensitivity to any of the components of oxaliplatin or pemetrexed
* Received radiotherapy to more than 25% of their bone marrow, or patients who received any radiotherapy within 4 weeks of entry
* Received treatment with strontium
* Receiving concurrent investigational therapy or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment
* Life expectancy < 6 months
* Peripheral neuropathy >= Grade 2
* Any other medical condition, including mental illness or substance abuse
* History of allogeneic transplant
* Known human immunodeficiency virus (HIV) or Hepatitis B or C (active, previously treated, or both)
* Inability to stop nonsteroidal anti-inflammatory drugs (NSAIDS) for a period of 2 days before, the day of, and 2 days following administration of Alimta; 5 days before, the day of, and 2 days following administration of Alimta for long-acting NSAIDS

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-06; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Pinski, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Dorff TB, Tsao-Wei DD, Groshen S, Boswell W, Goldkorn A, Xiong S, Quinn DI, Pinski JK. Efficacy of oxaliplatin plus pemetrexed in chemotherapy pretreated metastatic castration-resistant prostate cancer. Clin Genitourin Cancer. 2013 Dec;11(4):416-22. doi: 10.1016/j.clgc.2013.07.011. Epub 2013 Oct 4. PMID 24099865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on June 14, 2006 and was closed to accrual on May 11, 2009 after accruing 47 subjects. Participants were recruited at LAC+USC Medical Center and the USC/Norris Cancer Hospital.
Pre-assignment Details: The study had no pre-assignment criteria.
Period: Overall Study
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor)
Started | 47
Completed | 43
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor)
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: For patients with measurable disease, the RECIST 1.0 criteria was used to determine response. Complete Response = disappearance of all target lesions, Partial Response = greater or equal to 30% decrease in sum of longest diameter or target lesions, Stable Disease = <30% decrease or <20% increase, Progressive Disease = greater or equal to 20% increase in longest diameter of target lesions. For patients who do not have measurable disease by RECIST, the response was based on PSA response defined by Prostate Cancer Working Group criteria (1999) as 50% reduction in PSA confirmed on a second measurement at least 4 weeks later.
Time Frame: RECIST evaluation: Baseline, after every 2 courses, and then every 6 months after off-study, up to 1 year. PSA evaluation: baseline, day 1 of each course, final evaluation, and then every 6 months after off-study, up to 1 year
Population: All participants who received at least 1 cycle of treatment were included.
Measure: Number; unit: Participants
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor)
Number analyzed (Participants) | 47
Participants
  Complete Response | 0
  Partial Response | 14
  Stable Disease | 21
  Progressive Disease | 8
  Inevaluable | 4

2. Secondary Outcome: Time to Disease Progression and Overall Survival
Description: Progression-free survival was defined as the time from the first infusion of study treatment to the date of radiographic disease progression according to RECIST 1.0, or until two consecutive PSA rises occurred with an absolute increase of 5 ng/mL and a 50% relative increase over baseline. For patients without documented disease progression, the date of death or last follow-up without disease progression was used.
Time Frame: Baseline, after every 2 courses, and then every 6 months after off-study (RECIST) until progression; or baseline, day 1 of each course, at the final evaluation, and then every 6 months after off-study (PSA) until progression
Population: Participants who received at least the first infusion of treatment were included.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor)
Number analyzed (Participants) | 47
Months
  Median Survival | 12.0 [9.8 to 17.2]
  Median Time to Progression | 5.8 [3.9 to 8.1]
  Median Progression Free Survival | 5.4 [3.8 to 6.9]

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Safety evaluation according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: Baseline, days 1 and 7 of each course, and at last evaluation, up to 1 year
Population: All participants who started treatment were included.
Measure: Number; unit: Participants
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor)
Number analyzed (Participants) | 47
Participants | 35

ADVERSE EVENTS:
Time Frame: Baseline, days 1 and 7 of each course, and at last evaluation
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor)
Serious Adverse Events (participants affected / at risk) | 35/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy and Enzyme Inhibitor) (N=47)
Alkaline Phosphatase (Investigations) | 5 (9)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 3 (3)
Death not associated with CTCAE term (Disease progression NOS) (General disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (4)
Dyspsnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 7 (7)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6 (6)
Hemoglobin (Blood and lymphatic system disorders) | 6 (8)
Infection - Other (Infections and infestations) | 1 (1)
Infection (documented clinically or microbiologically) with Gr 3 or 4 neutrophis (ANC <1.0 x 10e9/L) (Infections and infestations) | 1 (1)
Infection with normal ANC or Gr 1 or 2 neutrophils (Blood) (Infections and infestations) | 1 (1)
Infection with normal ANC or Gr 1 or 2 neutrophils (Upper airway NOS) (Infections and infestations) | 1 (1)
Leukocytes (total WBC) (Investigations) | 7 (10)
Lymphopenia (Investigations) | 9 (20)
Muscle weakness, generalized or specific area (not due to neuropathy) (Whole body/generalized) (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 9 (25)
Pain (Back) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Bone) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Extremity-limb) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Joint) (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain (Muscle) (Musculoskeletal and connective tissue disorders) | 6 (6)
Platelets (Investigations) | 2 (3)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy and Enzyme Inhibitor) (N=47)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 19 (41)
Alkaline Phosphatase (Investigations) | 39 (69)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 14 (18)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 20 (33)
Anorexia (Metabolism and nutrition disorders) | 35 (71)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 35 (64)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (5)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 3 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 9 (12)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 11 (13)
Constitutional Symptoms (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine Increased (Investigations) | 12 (24)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 17 (35)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 20 (24)
Dry eye syndrome (Eye disorders) | 1 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 (2)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Edema: limb (General disorders) | 7 (9)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 47 (129)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (3)
Flu-like syndrome (General disorders) | 4 (4)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 36 (76)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 10 (10)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 10 (16)
Hemoglobin-decreased (Blood and lymphatic system disorders) | 47 (103)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Incontinence, anal (Gastrointestinal disorders) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Bladder [urinary]) (Infections and infestations) | 2 (2)
Infection with unknown ANC (Bladder [urinary]) (Infections and infestations) | 1 (1)
Injection site reaction/extravasation changes (General disorders) | 2 (2)
Leucocytes (total WBC)-decreased (Investigations) | 29 (95)
Lymphopenia (Investigations) | 3 (3)
Memory impairment (Nervous system disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Whole body/generalized) (Musculoskeletal and connective tissue disorders) | 3 (3)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (3)
Nasal cavity/paranasal sinus reactions (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 31 (53)
Neuropathy: cranial (CN VIII Hearing and balance) (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 40 (87)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 24 (43)
Pain (Abdomen NOS) (Gastrointestinal disorders) | 4 (5)
Pain (Back) (Musculoskeletal and connective tissue disorders) | 7 (8)
Pain (Bone) (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (Chest/thorax NOS) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Extremity-limb) (Musculoskeletal and connective tissue disorders) | 7 (9)
Pain (Head/headache) (Nervous system disorders) | 2 (2)
Pain (Joint) (Musculoskeletal and connective tissue disorders) | 29 (51)
Pain (Muscle) (Musculoskeletal and connective tissue disorders) | 29 (45)
Pain (Oral cavity) (Gastrointestinal disorders) | 1 (1)
Pain (Stomach) (Gastrointestinal disorders) | 2 (2)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 7 (11)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 5 (5)
Platelet count decreased (Investigations) | 19 (58)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 6 (8)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (4)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 25 (36)
Supraventricular and nodal arrhythmia (Sinus tachycardia) (Cardiac disorders) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1)
Taste alteration (dysgeusia) (Nervous system disorders) | 3 (3)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 5 (7)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 16 (21)
Watery eye (epiphora, tearing) (Eye disorders) | 1 (1)
Weight loss (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes